CLINICAL TRIAL: NCT01843504
Title: The Clinical, Biomechanical, and Tissue Regenerating Effects of a Single Platelet-rich Plasma Injection for the Treatment of Chronic Patellar Tendinopathy: a Randomized Controlled Trial
Brief Title: Platelet-Rich Plasma (PRP) Injection for the Treatment of Chronic Patellar Tendinopathy
Acronym: PRP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0177; 2012-0723 (Other: UW IRB); Protocol Version Date 1/29/16 (Other: UW Madison)
Record Dates: First submitted 2013-04-25; First posted 2013-04-30 (Estimated); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Chronic Patellar Tendinopathy; Chronic PT
Keywords: platelet rich plasma; PRP; plasma; plasma injection; patellar tendinopathy; patella tendon; patella; ultrasound; shear wave ultrasound; tendinosis; tendinopathy; tendinitis; jumper's knee
MeSH Terms: conditions — Patella Fracture; Tendinopathy | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma (Active Comparator): Subjects in Group 1 (PRP) will receive a single US-guided injection of 5 mL autologous platelet-rich plasma at week 0 (baseline).
  Interventions: Biological: platelet rich plasma
- Group 2 (Placebo Comparator): Subjects in Group 2 (saline control) will receive a single injection of 5 mL 0.9% normal saline at week 0.
  Interventions: Other: saline

INTERVENTIONS:
Biological: platelet rich plasma — A blood draw of 15 mL of the subject's own blood will be performed. The study coordinator will then place the sample in the Platelet Separator System (a centrifuge) and spin the blood sample in using a two-stage spinning: the 1st separates red blood cells from platelets, and the 2nd concentrates the platelets. This will be spun by centrifuge to yield 6 mL of concentrated autologous platelet. Under continuous ultrasound evaluation, 1.0-2.0 mL of the prepared PRP will be injected onto the origin of the patella tendon itself will be peppered along a short segment of the tendon into the areas of palpated tenderness and US-documented pathology.
  Arms: Platelet Rich Plasma
Other: saline — A blood draw of 15 mL of the subject's own blood will be performed to maintain blinding. Under continuous ultrasound evaluation, 1.0-2.0 mL of the saline solution will be injected onto the origin of the patella tendon itself will be peppered along a short segment of the tendon into the areas of palpated tenderness and US-documented pathology.
  Arms: Group 2

SUMMARY:
The goal of this study is to find an effective treatment for chronic patellar tendinopathy (PT). Investigators will conduct a 32-week randomized controlled clinical trial to determine whether platelet rich plasma (PRP) injections improve disease-specific clinical outcomes with correlation to a new method of ultrasound (US) imaging assessment called Acoustoelastography (AE). Positive findings of PRP compared to control would suggest future larger scale studies to help establish an optimal protocol for the nonsurgical management of PT.

DETAILED DESCRIPTION:
This study is a randomized, single-blinded controlled trial. Subjects, aged 18-65 with chronic patellar tendinopathy (PT), will be recruited through the University of Wisconsin (UW) Sports Medicine Clinics and the UW Physical Therapy Clinics. 44 subjects will be randomized to one of two study arms (22 in each group). Subjects and assessors will be blinded to the subject group allocation.

Subjects in Group 1 (PRP) will receive a single US-guided injection of up to 5 mL autologous platelet-rich plasma at week 0 (baseline). Subjects in Group 2 (saline control) will receive a single injection of 5 mL 0.9% normal saline at week 0. Subjects in both groups will receive just one session of injection.

Subjects invited to participate in the study will be asked to undergo a knee evaluation examination. Tender areas associated with the patellar tendon will be identified. This exam will occur at the US Sports Medicine Clinic at Research Park. If patient is being seen by PI for a routine clinic visit for knee pain, patient may be identified as a potential research participant. During the clinic visit, the patient will undergo a knee evaluation examination. If patient is confirmed to have patellar tendinopathy, the PI will introduce the study. If interested, the PI will conduct a brief in-person interview to determine eligibility via self-reported inclusion and exclusion criteria. Subjects who qualify will have written consent obtained prior to their knee exam.

Subjects will then report to WIMR where the ultrasound-guided procedures and follow-up diagnostic imaging will be conducted. The study coordinator will greet the subjects, remind them of the details of the study procedure, its potential benefits and risks, and answer questions. Dr. Lee will then meet the subject, answer any questions and assess vital signs.

The RN will prepare a 3 mL syringe of 1% lidocaine with a 30G, ½" long needle for pre-injection topical analgesia (skin wheal).

The RN will then perform a blood draw of 15 mL of the subject's own blood from the antecubital fossa of the elbow using a 20 mL syringe and an 18G needle. There is no side preference. Control subjects will also undergo phlebotomy to maintain blinding. This is a small amount of blood; Red Cross donations of one unit of whole blood are typically 450 mL. The study coordinator will then place the sample in the Platelet Separator System (a centrifuge) and spin the blood sample in using a two-stage spinning: the 1st separates red blood cells from platelets, and the 2nd concentrates the platelets. This will be spun by centrifuge to yield 6 mL of concentrated autologous platelet. All blood and equipment handling will follow universal precautions.

Ultrasound will serve as visual guidance for injections. Dr. Lee will perform all ultrasound-guided injections. The injection technique is identical for subjects in the two injection groups. The skin will be cleansed with chloraprep. Lidocaine skin wheals will be placed for local analgesia. The origin of the patellar tendon of the affected knee will be identified using the ultrasound12MHz linear array transducer. Under continuous ultrasound evaluation, 1.0-2.0 mL of the prepared PRP or saline solution will be injected onto the origin of the patella tendon itself using a 22G, 1.5" long needle. Then, 3.0 to 4.0 mL of the PRP or saline solution will be peppered along a short segment of the tendon into the areas of palpated tenderness and US-documented pathology.

Ultrasound guided PRP injections and follow-up ultrasound will be performed at WIMR's Ultrasound Imaging Research Lab. The WIMR Ultrasound research program will provide the equipment (Siemens S2000), linear array probes, and supplies for injections. The WIMR Ultrasound research program will provide the research sonographer (Sarah Kohn). This is important in maintaining consistency in imaging protocol, image acquisition, and subject satisfaction, which also influences outcomes of research studies.

After the injections, the subjects will rest for 5 minutes and the study coordinator will then obtain the subject's vital signs. Subjects will be asked to complete outcome questionnaires. Participants will be given 20 tablets of 500mg acetaminophen for "as-needed" analgesia and will be telephoned after 2 days to enquire about side effects or adverse events outcome assessment procedures.

The platelet concentration will be analyzed in both samples (whole blood compared to PRP) in order to verify the concentration factor in PRP. Platelet counts in whole blood vary by individual. The optimal quantity of platelets and growth factors required for tissue healing is not known, but a clinically effective concentration has been described as being greater than 4 times baseline autologous whole blood platelet concentrations. Therefore, platelet concentration yield may have important implications in clinical outcome correlation.

Following the procedure, approximately 1 mL of autologous whole blood and 1 mL of unused PRP will be analyzed using a standard lab automated analyzer, a Horiba ABX Micros 60 hematology cytometer, at the UW Health Research Park Clinic.

Subjects will complete outcome questionnaires at weeks 0, 4, 8, 12, 16, and 32 weeks. The questionnaires for weeks 4, 8, 12 and 16, along with self-addressed stamped envelopes will be provided to study participants at the time of enrollment in their study folder. Questionnaires will be returned at the time of the indicated due date at the top of the questionnaires. If subjects do not return their questionnaires, a member of the study team will contact the subjects by phone as a reminder, and the participant will be invited to complete the survey by phone.

Ultrasound imaging will be performed at baseline and 32 weeks. On the final visit, participants will report for a scheduled visit to the WIMR clinic for their 32 week ultrasound visit. Subjects will complete their 32 week questionnaires at that time if subjects have not already done so.

ELIGIBILITY:
Inclusion Criteria:

1. age18-65
2. chronic (>3months) patellar tendon pain;
3. clinical exam findings consistent with PT;
4. self-reported failure of supervised physical therapy;
5. self-reported failure of at least 2 of the most common treatments (NSAIDs, relative rest, ice, bracing) for patellar tendinopathy.

Exclusion Criteria:

1. inability to comply with follow-up requirements of study,
2. history of bleeding disorders, low-platelet counts, other hematologic conditions;
3. knee pain due to another possible etiology(e.g., degenerative joint disease);
4. current or recent use of anticoagulation or immunosuppressive therapy;
5. known allergy to acetaminophen or Lidocaine;
6. self-reported pregnancy;
7. worker's compensation injury;
8. pending litigation;
9. concurrent opioid use for pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change in Victorian Institute of Sport Assessment-Patellar (VISAP) Score | 0, 4, 8, 12, 16, and 32 weeks
  Participants will complete outcome questionnaires at weeks 0, 4, 8, 12, 16, and 32 weeks. The results will evaluate pain- and function-dependent, knee-specific quality of life, as assessed by composite scores on the validated Victorian Institute of Sport Assessment-Patellar (VISAP). The total possible range of scores is 0-100 with higher scores indicating fewer symptoms and higher function.
Change in International Knee Documentation Committee (IKDC) Score | 0, 4, 8, 12, 16, and 32 weeks
  Participants will complete outcome questionnaires at weeks 0, 4, 8, 12, 16, and 32 weeks. The results will evaluate pain- and function-dependent, knee-specific quality of life, as assessed by composite scores on the International Knee Documentation Committee (IKDC). The total possible range of scores is 0-100 with higher scores indicating increased discomfort and interference with daily activities.
Change in Knee Injection Questionnaire Score | 0, 4, 8, 12, 16, and 32 weeks
  Participants will complete outcome questionnaires at weeks 0, 4, 8, 12, 16, and 32 weeks. The results will evaluate pain- and function-dependent, knee-specific quality of life, as assessed by composite scores on the Knee Injection Questionnaire. The total possible range of scores is 0-100 with higher scores indicating improved well being and ability to activities.

SECONDARY OUTCOMES:
Change in Thickness of Patellar Tendon Compared to Contralateral | baseline to 32 weeks
  Ultrasound (US) changes of several pathologic features of PT will be evaluated using US imaging of the patellar tendon at 32 weeks compared to baseline imaging. Conventional ultrasound will be done to assess patellar tendon thickness (contralateral comparison).
Change in Neovascularity of Patellar Tendon | baseline to 32 weeks
  Ultrasound (US) changes of several pathologic features of PT will be evaluated using US imaging of the patellar tendon at 32 weeks compared to baseline imaging. Conventional ultrasound will be done to assess patellar tendon neovascularity.
Change in Hypoechogenicity of Patellar Tendon | baseline to 32 weeks
  Ultrasound (US) changes of several pathologic features of PT will be evaluated using US imaging of the patellar tendon at 32 weeks compared to baseline imaging. Conventional ultrasound will be done to assess patellar hypoechogenicity.
Change in Stiffness of Patellar Tendon | baseline to 32 weeks
  Acoustoelastography (AE) will be done to measure stiffness changes of the patellar tendon using standardized 0-3 severity scales compared to control subjects.

OTHER OUTCOMES:
Knee Injection Survey: PRP Satisfaction Questionnaire | up to 32 weeks
  Outcome measures will be compared for satisfaction with PRP therapy as assessed by the treatment satisfaction survey score at 32 weeks post-treatment. This survey is a 5-item survey that assesses
  * severity of symptoms (0 no symptoms to 6 worst symptoms)
  * level of difficulty in using the knee, if any, (1 mild to 4 unable to use knee)
  * change in knee symptoms since treatment (-3 very much worse to 0 no change to 3 very much improved)
  * physical ease, comfort, convenience, and effectiveness satisfaction with PRP therapy (each from -3 extremely dissatisfied to 0 neutral to 3 extremely satisfied), and
  * temporary pain, bruising, swelling, bleeding, or other side effects (from 5 all of the time to 0 none of the time)

CONTACTS AND LOCATIONS:
Overall Officials: John J. Wilson, MD, MS, Principal Investigator — UW-Madison School of Medicine & Public Health; Stephen J. Almasi, MD, Principal Investigator — UW-Madison School of Medicine & Public Health; Kenneth S. Lee, MD, Principal Investigator — UW-Madison School of Medicine & Public Health
Locations (2):
- United States (2):
  - Wisconsin Institute of Medical Research, Madison, Wisconsin
  - UW Sports Medicine Clinic at Research Park, Madison, Wisconsin

REFERENCES:
- [Background] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519